CLINICAL TRIAL: NCT02120599
Title: Randomized Controlled Trial of the Impact of Treating Moderately Malnourished Women in Pregnancy
Brief Title: Interventions for Moderate Malnutrition in Pregnancy
Acronym: Mamachiponde
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201401112
Record Dates: First submitted 2014-04-18; First posted 2014-04-23 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Pregnancy; Moderate Malnutrition
MeSH Terms: interventions — Iron; Folic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- corn-soy-blend (Active Comparator): This is the control group for the study, which will receive the Malawi standard of care. The treatment provided to women randomized to this arm of the study includes daily iron (60 mg) and folic acid (400 mcg) supplementation, along with 4 kg/2 weeks corn-soy blend (~357 gm/d CSB).
  Interventions: Dietary Supplement: corn-soy blend; Dietary Supplement: iron; Dietary Supplement: folic acid
- corn-soy-blend + multiple micronutrients (Experimental): The treatment provided to women randomized to this arm of the study includes 200gm/d CSB along with a standard maternal multiple micronutrient tablet, which together provide a comparable amount of energy, protein and micronutrients to the ready-to-use supplemental food. The micronutrient supplement known as the United Nations Children's Emergency Fund (UNICEF) / World Health Organization (WHO) / United Nations University (UNU) international multiple micronutrient preparation (UNIMMAP) is widely available and has been used in many settings worldwide in pregnant women.
  Interventions: Dietary Supplement: corn-soy blend; Dietary Supplement: UNIMMAP
- ready-to-use supplementary food (Experimental): RUSF-P (ready-to-use supplementary food) provides 750 kcal/d, 20 g protein/d, and 200% of RDA/d for most micronutrients during pregnancy (except for vitamins A, B3, folic acid, minerals iodine, magnesium, and calcium which will remain near 100%)
  Interventions: Dietary Supplement: ready-to-use supplementary food

INTERVENTIONS:
Dietary Supplement: ready-to-use supplementary food
  Arms: ready-to-use supplementary food
Dietary Supplement: corn-soy blend
  Arms: corn-soy-blend; corn-soy-blend + multiple micronutrients
Dietary Supplement: iron
  Arms: corn-soy-blend
Dietary Supplement: folic acid
  Arms: corn-soy-blend
Dietary Supplement: UNIMMAP
  Arms: corn-soy-blend + multiple micronutrients

SUMMARY:
Malnutrition during pregnancy is more common in poor women in the developing world due to inadequate dietary intake combined with increased nutrient requirements; pregnancy risk is more consequential than among other demographic groups with increased risk of maternal and infant mortality and the lifelong effects of fetal malnutrition. The benefits of treating moderate malnutrition during pregnancy remain largely undocumented. This study tests the hypothesis that providing either a fortified flour or fortified paste-based supplementary food designed to replete the nutrient deficits during pregnancy will result in improved maternal nutritional recovery rates and higher infant birth weights and lengths. This study is a randomized, controlled clinical trial of 3 supplementary foods in 1800 moderately malnourished Malawian women who are pregnant. Subjects will receive one of 3 food rations: 1) a ready-to-use supplementary food formulated to deliver about 200% of the recommended daily allowance (RDA) of most micronutrients in pregnancy (RUSF-P), 2) corn soy blend with a multiple micronutrient tablet chosen to deliver about 200% of the RDA of most micronutrients (CSB-P) or 3), the standard of care which is a corn soy blend with supplementary iron and folic acid (CSB), delivering between 0-350% of the RDA. Subjects will receive the supplementary food until they recover from MAM. The outcome of the pregnancy and maternal nutritional status will be followed until 3 months after delivery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and consenting to study participation and HIV testing (if not already performed)
* mid-upper-arm circumference (MUAC) ≤ 23 cm
* planning to stay in the area and attend the clinic during pregnancy and for 3 months post partum

Exclusion Criteria:

* Pregnancy complications such as gestational diabetes, pre-eclampsia, hypertension
* Severe anemia (Hg <7.0 mg/dl)
* Severe malnutrition
* under 18 years of age
* over estimated 35 weeks of gestation

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1867 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Proportion recovered from moderate acute malnutrition (MAM) | up to 40 weeks
  proportion of women who reach mid-upper arm circumference (MUAC) > 23.5 cm for 2 consecutive visits
Maternal change in mid-upper arm circumference (MUAC) | up to 40 weeks
  average change in mid-upper-arm circumference
infant birth weight | up to 40 weeks
  mean birth weights of infants born to mothers in the study
infant birth length | up to 40 weeks
  mean birth length of infants born to women in the study
premature delivery | up to 36 weeks
  proportion of infants born prematurely

SECONDARY OUTCOMES:
maternal weight gain | up to 40 weeks
maternal hemoglobin | 8 weeks
  changes in average hemoglobin level
pregnancy complications | up to 40 weeks
  rate of pregnancy complications
infant weight at 3 months | 3 months
infant length at 3 months | 3 months
infant survival at 3 months | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Manary, MD, Study Chair — Washington University in St. Louis; University of Malawi; Peggy C Papathakis, PhD, RD, Study Director — California Polytechnic State University-San Luis Obispo; Kenneth Maleta, MBBS PhD, Principal Investigator — University of Malawi; Chrissie Thakwalakwa, Principal Investigator — University of Malawi
Locations (2):
- Malawi (2):
  - Blantyre District, Blantyre
  - Chikwawa District, Chikwawa

REFERENCES:
- [Derived] Callaghan-Gillespie M, Schaffner AA, Garcia P, Fry J, Eckert R, Malek S, Trehan I, Thakwalakwa C, Maleta KM, Manary MJ, Papathakis PC. Trial of ready-to-use supplemental food and corn-soy blend in pregnant Malawian women with moderate malnutrition: a randomized controlled clinical trial. Am J Clin Nutr. 2017 Oct 1;106(4):1062-1069. doi: 10.3945/ajcn.117.157198. PMID 28793991